CLINICAL TRIAL: NCT05979688
Title: Yogic Breathing Exercise for People With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hon K. Yuen, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300011535
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis; Myasthenia Gravis
Keywords: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors are masked to participant group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yogic breathing exercise (Experimental): Participation in a 6 weekly virtual yogic breathing exercise training with 1-3 sessions per week.
  Interventions: Behavioral: yogic breathing exercise
- Waitlist control (No Intervention): Participation in usual daily activities

INTERVENTIONS:
Behavioral: yogic breathing exercise — A typical session will begin with the yoga instructor demonstrating a breathing exercise technique. The participants will learn and practice each technique.
  Arms: Yogic breathing exercise

SUMMARY:
The aim of this study is to understand how well a 6-week virtual yogic breathing exercise program (YBEP) will improve breathing, speech, and emotional well-being in people with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
The study will employ a RCT to test the two hypotheses. The study will incorporate a 2 x 2 two-way factorial design with repeated measures at three time points. The two between-subject factor conditions will be participation in a yogic breathing exercise program (YBEP) versus a waitlist control condition that will be evaluated at baseline, and immediately post-program. Thirty adults with ALS will be recruited for this study.

Hypothesis #1: Adults with ALS who participate in a YBEP will demonstrate improvement in breathing, and emotional well-being compared to waitlist controls at the conclusion of a 6-week YBEP.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed ALS or myasthenia gravis diagnosis
2. age >18 yrs old;
3. ability to follow multistep commands,
4. on a stable dose of medications for >60 days,
5. FVC ≥30% predicted,
6. access to internet and a computer or smartphone that can perform videoconferencing.

Exclusion Criteria:

1. life expectancy is less than 6 months,
2. severe hearing or visual impairments that prevent online learning (breathing exercise), or
3. current participation in another clinical trial during the study period that can affect the outcomes of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
ALS Specific Quality of Life-Revised | baseline
  ALS Specific Quality of Life-Revised (ALSSQOL-R) consists of 6 subscales: negative emotion (13 items), interaction with people and the environment (11 items), intimacy (7 items), religiosity (4 items), physical symptoms (6 items), and bulbar function (5 items). The scale has 46 items rated on a 11-point Likert-type scale (0 to 10) with higher scores indicating better quality of life. Some items require reverse scoring.
ALS Specific Quality of Life-Revised | at 6 weeks
  ALS Specific Quality of Life-Revised (ALSSQOL-R) consists of 6 subscales: negative emotion (13 items), interaction with people and the environment (11 items), intimacy (7 items), religiosity (4 items), physical symptoms (6 items), and bulbar function (5 items). The scale has 46 items rated on a 11-point Likert-type scale (0 to 10) with higher scores indicating better quality of life. Some items require reverse scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Hon Yuen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pagnini F, Marconi A, Tagliaferri A, Manzoni GM, Gatto R, Fabiani V, Gragnano G, Rossi G, Volpato E, Banfi P, Palmieri A, Graziano F, Castelnuovo G, Corbo M, Molinari E, Riva N, Sansone V, Lunetta C. Meditation training for people with amyotrophic lateral sclerosis: a randomized clinical trial. Eur J Neurol. 2017 Apr;24(4):578-586. doi: 10.1111/ene.13246. Epub 2017 Feb 23. PMID 28229508